CLINICAL TRIAL: NCT00524576
Title: Administration of a Challenge Dose of Hepatitis B Vaccine in Subjects Who Previously Received Engerix™-B Vaccine.
Brief Title: Challenge Dose of Hepatitis B Vaccine in Subjects Who Previously Received Engerix™-B Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 108988
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Persistence; Challenge dose
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

ARMS (2):
- Engerix 2 Doses + Challenge Dose (Experimental): Subjects received 2 doses of Engerix™-B (Month 0 and 6) in the primary study and a single dose of Engerix™-B during the booster study.
  Interventions: Biological: Engerix™-B
- Engerix 3 Doses + Challenge Dose (Experimental): Subjects received 3 doses of Engerix™-B (Month 0, 1 and 6) in the primary study and a single dose of Engerix™-B during the booster study.
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Engerix™-B — One dose (10µg Hepatitis B surface antigen (HBsAg))
  Other Names: Hepatitis B vaccine

SUMMARY:
To evaluate the response to an additional dose (challenge dose) of hepatitis B vaccine, when given to subjects who had received primary vaccination of Engerix™-B vaccine approximately 72-78 months ago.

This protocol posting deals with objectives & outcome measures of the challenge phase. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female who had received complete primary vaccination course of hepatitis B vaccine in the primary study
* Written informed consent obtained from the subject and/or parent/guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after the hepatitis B challenge dose.

Exclusion Criteria:

* Use of any investigational/non-registered drug or vaccine other than the study vaccine within 30 days preceding the hepatitis B vaccine challenge dose or planned use during the study period.
* Chronic administration (more than 14 days) of immunosuppressants other immune-modifying drugs within six months prior to the hepatitis B vaccine challenge dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before the hepatitis B vaccine challenge dose and ending 30 days after.
* Subjects who received an additional dose of hepatitis B vaccine outside the context of the study between the primary vaccination course and the hepatitis B challenge vaccination visit.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the hepatitis B vaccine challenge dose or planned administration during the study period (one month).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2007-11-28; Primary Completion 2008-05-14 (Actual); Study Completion 2008-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Westmead, New South Wales, Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Damme P, Moiseeva A, Marichev I, Kervyn AD, Booy R, Kuriyakose S, Brockway A, Ng SP, Leyssen M, Jacquet JM. Five years follow-up following two or three doses of a hepatitis B vaccine in adolescents aged 11-15 years: a randomised controlled study. BMC Infect Dis. 2010 Dec 20;10:357. doi: 10.1186/1471-2334-10-357. PMID 21171982
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 108988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108988 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Started | 97 | 47
Completed | 97 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose | Total
Number analyzed (Participants) | 97 | 47 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (1.22) | 19.3 (1.46) | 19.4 (1.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 23 | 73
  Male | 47 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immunological Response to Challenge Dose in Terms of Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration
Description: Immune response defined as:
  * For initially seronegative subjects (anti-HBs antibody concentration <3.3 milli-international unit per milliliter [mIU/mL] before vaccination) antibody concentration ≥ 10mIU/mL at post booster.
  * For initially seropositive subjects: antibody concentration at post booster ≥ 4-fold the pre-vaccination antibody concentration.
Time Frame: 30 days post-challenge dose
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity. Data from the Australian center were not included following data quality issues detected at the investigator site.
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 53 | 21
participants | 53 | 21

2. Secondary Outcome: Number of Participants With Anti-HBs Antibody Concentrations Above the Cut-off Value
Description: Anti-HBs antibody cut-off values assessed include 3.3, 10 and 100 mIU/mL.
Time Frame: 30 days post-challenge dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 53 | 21
participants
  ≥ 3.3 mIU/mL | 53 | 21
  ≥ 10 mIU/mL | 53 | 21
  ≥ 100 mIU/mL | 50 | 20

3. Secondary Outcome: Concentration of Anti-HBs Antibodies
Description: Concentrations given as geometric mean concentration (GMC) and expressed in mIU/mL.
Time Frame: 30 days post-challenge dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 53 | 21
mIU/mL | 6214.1 [3213.1 to 12018.0] | 16564.3 [6394.9 to 42905.6]

4. Secondary Outcome: Number of Participants Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 4-day follow-up period (Day 0-3) after the challenge dose
Population: Analysis was performed on the Total Vaccinated Cohort. Data from the Australian center were not included following data quality issues detected at the investigator site.
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 55 | 22
participants
  Pain | 22 | 4
  Redness | 11 | 1
  Swelling | 9 | 0

5. Secondary Outcome: Number of Participants Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include fatigue, fever, gastrointestinal symptoms, and headache.
Time Frame: During the 4-day follow-up period (Day 0-3) after the challenge dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 55 | 22
participants
  Fatigue | 19 | 7
  Fever ≥ 37.5 degree Celsius | 1 | 0
  Gastrointestinal disorder | 7 | 4
  Headache | 14 | 4

6. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day follow-up period (Day 0-30) after the challenge dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 55 | 22
participants | 19 | 5

7. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 31-day follow-up period (Day 0-30) after the challenge dose
Population: Analysis was performed on the Total Vaccinated Cohort. This table describes SAEs reported by all subjects except for those enrolled in the Australian center.
Measure: Number; unit: participants
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
Number analyzed (Participants) | 55 | 22
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day follow-up period (Day 0-3) after the challenge dose. Unsolicited AEs and serious AEs (SAEs): during the 31-day follow-up period (Day 0-30) after the challenge dose.
Description: Data from the Australian center were not included following data quality issues detected at the investigator site.
Arm/Group | Engerix 2 Doses + Challenge Dose | Engerix 3 Doses + Challenge Dose
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/22
Other Adverse Events (participants affected / at risk) | 39/55 | 14/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engerix 2 Doses + Challenge Dose (N=55) | Engerix 3 Doses + Challenge Dose (N=22)
Headache (Nervous system disorders) | 17 (18) | 6 (6)
Pain (General disorders) | 22 (22) | 4 (4)
Redness (General disorders) | 11 (11) | 1 (1)
Swelling (General disorders) | 9 (9) | 0 (0)
Fatigue (General disorders) | 19 (19) | 7 (7)
Gastrointestinal disorder (General disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.